CLINICAL TRIAL: NCT05803057
Title: Beijing Neurosurgical Institute, Beijing, China
Brief Title: Accelerating Motor Recovering in Patients With SMA Syndrome After Glioma Surgery by Using nrTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Principal Investigator, TAO JIANG, Director, Department of Neurosurgery, Principal Investigator, Clinical Professor, Beijing Neurosurgical Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8220101798
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Motor Cortex; Lesion; Glioma; Supplementary Motor Area Syndrome
Keywords: human; motor recovery; transcranial magnetic stimulation
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: There are two groups of this study. The one is that the patients receive nrTMS stimulation with high-frequency on the thumb-related motor cortex on the lesional hemisphere. The other is that the patients receive nrTMS sham-stimulation with high-frequency on the thumb-related motor cortex on the lesional hemisphere.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There are two stimulating colis with the same shape, color and touch. The one is able to stimulate, the other is able to sham-stimulate. All patients are randomly assigned to use one of the two coils for treatment. Except for the designer, all participant, care provider, investigator, and outcomes assessorthey don not know who used which coil to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS treatment (Experimental): Using nrTMS coli to stimulate the thumb related motor cortex with high-frequency.
  Interventions: Device: TMS stimulation treatment
- TMS Sham-treatment (Sham Comparator): Using nrTMS sham-coli to stimulate the thumb related motor cortex with high-frequency.
  Interventions: Device: TMS stimulation sham-treatment

INTERVENTIONS:
Device: TMS stimulation treatment — Using the TMS treatment coli to stimulation with high frequency
  Arms: TMS treatment
Device: TMS stimulation sham-treatment — Using the TMS sham-treatment coli to stimulation with high frequency
  Arms: TMS Sham-treatment

SUMMARY:
The goal of this randomized clinical controlled trial is to learn about whether neuro-navigation repetitive transcranial magnetic stimulation (nrTMS) was useful to accelerate the recovery in patients with SMA syndrome after glioma resection. The main questions aim to answer:

* Question 1: Whether the nrTMS was useful to accelerate the recovery of motor function back to the preoperative status in participants with SMA syndrome after glioma resection.
* Question 2: Whether the nrTMS was useful to improve postoperative motor function in participants with SMA syndrome after glioma resection.

Participants will continue to receive nrTMS treatment or nrTMS sham-treatment for 7 times on the 8th day after glioma resection to determine whether the TMS was helpful for exercise rehabilitation. The investigator will evaluate the effects of nrTMS treatment through the ratio of recovery of motor function and the time that was from the participants suffering SMA syndrome to totally recover the motor function to the status of motor function in pre-operation.

DETAILED DESCRIPTION:
This study will use the 8-coil (Magstem, England, No.4150) and sham 8-coil (Magstem, England) The criteria of enrolled patients are： A. Inclusion time: from April 01 2023 to March 31 2025 (including the current month); B. Inpatients in neurosurgery oncology wards of Beijing Tiantan Hospital; C. Right-handed, age: 25-55 years old, tumor located in SMA, no previous treatment history of nervous system disease; D. The patient received wake-up surgery and applied direct cortical electrical stimulation during the operation to determine the location of the motor area; E. Postoperative pathology was low grade glioma; F. Can accept nrTMS rehabilitation treatment.

The excluding criteria are:

A. The tumor grows across the midline to the opposite side; B. When collecting rs-fMRI data, head movement exceeds 1mm and head deflection exceeds 1 °; C. The patient did not have SMA syndrome after operation; D. Vulnerable or special groups and protective measures, such as pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients in neurosurgery oncology wards of Beijing Tiantan Hospital
* Right-handed, age: 25-55 years old
* Tumor located in supplementary motor area
* No previous treatment history of central nervous system disease
* The patient received awaken craniotomy
* Pathological diagnosis is low grade glioma
* Volunteer to accept nrTMS treatment

Exclusion Criteria:

* The tumor grows across the midline to the opposite side
* Regarding rs-fMRI data, head movement exceeds 1mm and head deflection exceeds 1 °
* The patient did not have SMA syndrome after operation
* Vulnerable or special groups and protective measures, such as pregnant women

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Motor function totally recovering in evaluating with MRC (the UK Medical Research Council) muscle strength test | From the day of tumor resection to 3 months after tumor resection
  The motor function recovers back to the status in pre-operation. The motor status means that the muscle strength muscle of upper limb that is controlled by lesional hemisphere. Moreover, the recovering back means that the muscle strength achieves at grade 5 (healthy grade).

SECONDARY OUTCOMES:
Motor function improve in evaluating with MRC (the UK Medical Research Council) muscle strength test | From the day of tumor resection to 3 months after tumor resection
  The motor function improves compared with the day of SMA syndrome occuring. The motor status means that the strength muscle of upper limb that is controlled by lesional hemisphere. Moreover, the motor imporvement means that the muscle strength is higher than the SMA syndrome occurring but does not achieve grade 5 (healthy grade).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakajima R, Kinoshita M, Yahata T, Nakada M. Recovery time from supplementary motor area syndrome: relationship to postoperative day 7 paralysis and damage of the cingulum. J Neurosurg. 2019 Feb 8;132(3):865-874. doi: 10.3171/2018.10.JNS182391. Print 2020 Mar 1. PMID 30738403
- [Result] Fang S, Li L, Weng S, Zhang Z, Fan X, Jiang T, Wang Y. Increasing nodal vulnerability and nodal efficiency implied recovery time prolonging in patients with supplementary motor area syndrome. Hum Brain Mapp. 2022 Sep;43(13):3958-3969. doi: 10.1002/hbm.25896. Epub 2022 May 4. PMID 35507429